CLINICAL TRIAL: NCT07362563
Title: Effect of 3 Different Prebiotic Sodas on Postprandial Levels of GLP-1, PYY, Transit Time and Satiety Levels: An Acute, Randomized Controlled Pilot Study in Healthy Participants
Brief Title: Effect of Prebiotic Sodas on Postprandial Levels of GLP-1, PYY, Transit Time and Satiety Levels: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olipop, PBC (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: INQ-2534
Record Dates: First submitted 2026-01-09; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Satiety in Healthy Volunteers
MeSH Terms: interventions — sodium bicarbonate-based toothpaste

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Soda (Placebo Comparator): Participants will consume one 12 oz can of a control soda
  Interventions: Other: Control Soda
- Prebiotic Soda - Shelf Stable (Experimental): Participants will consume one 12 oz can of the shelf stable prebiotic soda
  Interventions: Other: Prebiotic Soda - Shelf Stable
- Prebiotic Soda - Refrigerated (Experimental): Participants will consume one 12 oz can of the refrigerated prebiotic soda
  Interventions: Other: Prebiotic Soda - Refrigerated
- Prebiotic Soda - Shelf Stable + Functional Ingredient (Experimental): Participants will consume one 12 oz can of the shelf stable prebiotic soda with an added functional ingredient
  Interventions: Other: Prebiotic Soda - Shelf Stable + Functional Ingredient

INTERVENTIONS:
Other: Control Soda — Participants will consume one 12 oz can of a control soda that contains 0 g dietary fiber and 4 g total sugar.
  Arms: Control Soda
Other: Prebiotic Soda - Shelf Stable — Participants will consume one 12 oz can of a shelf stable prebiotic soda that contains 6 g dietary fiber and 4 g total sugar.
  Arms: Prebiotic Soda - Shelf Stable
Other: Prebiotic Soda - Refrigerated — Participants will consume one 12 oz can of a shelf stable prebiotic soda that contains 9 g dietary fiber and 4 g total sugar.
  Arms: Prebiotic Soda - Refrigerated
Other: Prebiotic Soda - Shelf Stable + Functional Ingredient — Participants will consume one 12 oz can of a shelf stable prebiotic soda that contains 6 g dietary fiber, 4 g total sugar, and an added functional ingredient.
  Arms: Prebiotic Soda - Shelf Stable + Functional Ingredient

SUMMARY:
The main objective of this study is to evaluate the acute effects of prebiotic sodas on postprandial levels of glucagon-like peptide-1 (GLP-1), peptide YY (PYY), gastric emptying, and satiety levels in healthy adults.

DETAILED DESCRIPTION:
The primary aim of this clinical trial is to evaluate the effects of single-dose prebiotic sodas on on postprandial levels of GLP-1.

Participants (n=15) will be healthy males and healthy, non-pregnant, non-lactating females aged 18-60 years. Participants will consume a single dose of 3 different prebiotic sodas (6 - 9 g dietary fiber and 4 g total sugar per can) and one control soda (0 g dietary fiber and 4 g total sugar per can) in a randomized, crossover design over a period of 4-12 weeks with an interval of at least 1 week and at most 3 weeks between visits.

Secondary outcomes will include evaluating the effects of single-dose consumption of the control and prebiotic sodas on postprandial PYY, gastric emptying, and satiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years, inclusive.
* BMI between 18.0 and 30.0 kg/m2.
* Stable weight in the last 3 months (+/-5kg).
* Willing to abstain from unusual strenuous exercise, consuming alcoholic drinks and from taking fiber supplements for 24 hours before study days.
* Willing to refrain from smoking tobacco or e-cigarettes, and using marijuana in any form for 12h before and during study visits.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.
* Subjects must be eligible to receive income in Canada and be covered by a health insurance plan such as Ontario Health Insurance Plan (OHIP).

Exclusion Criteria:

* Self-reported pregnant or breastfeeding women.
* Subjects with a history of severe food allergies or an allergy to acetaminophen.
* Known history of diabetes, any gastrointestinal disorder that alters the absorption of nutrients, liver disease, or the presence of any health condition, illness or drug use that increases risk to the subject or to others or may affect the results, as judged by the Qualified Investigator (QI).
* Subjects who are currently or in the last 2 months have been on oral or injectable GLP-1 receptor agonist (RA) medications.
* Subjects who consume more than 14 alcoholic drinks per week, or more than 5 alcoholic drinks on any one occasion.
* Subjects who have been on antibiotic therapy in the last 2 months.
* Subjects taking the blood thinning drug warfarin.
* Subjects who are habitual users of the following supplements in the past 30 days: berberine, curcumin, cinnamon, resveratrol, and gardenia.
* Subjects which have undergone major surgery in the last 3 months.
* Unwillingness or inability to comply with experimental procedures and to follow Inquis safety guidelines.
* Subject is currently participating or recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement, or lifestyle modification.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Blood GLP-1 iAUC | For 2 hours post intervention
  Incremental area under the curve (iAUC) for GLP-1 from immediately prior to test-product consumption (t=0) to t=120 min following test-product consumption.

SECONDARY OUTCOMES:
Blood PYY iAUC | For 2 hours post intervention
  Incremental area under the curve (iAUC) for PYY from immediately prior to test-product consumption (t=0) to t=120 min following test-product consumption.
Gastric Emptying Rate/Transit Time via Acetaminophen | Oral dose of acetaminophen with blood samples taken for 2 hours post intervention
  Incremental area under the curve (iAUC) for acetaminophen from immediately prior to test-product consumption (t=0) to t=120 min following test-product consumption.
Change in Perceived Satiety Levels | For 2 hours post intervention
  The change in perceived satiety levels measured using the Motivation to Eat visual analogue scale (VAS) from immediately prior to test-product consumption (t=0) to t=120 min following test-product consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Campbell, Study Director — INQUIS Clinical Research
Locations (1):
- Inquis Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No